CLINICAL TRIAL: NCT05793255
Title: The Impact of Social Phone Calls on Adults Who Have Had a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jennifer Beauchamp, associate professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-22-1084
Record Dates: First submitted 2023-03-15; First posted 2023-03-31 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: stroke; phone calls; social support; loneliness; ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Behavioral: Social Phone Calls

INTERVENTIONS:
Behavioral: Social Phone Calls — Following the collection of baseline data, the study participant will be randomly assigned to a student volunteer to begin the social phone calls. The first phone call will be scheduled to occur within one week of the consent and baseline assessments. A minimum of one social phone call will occur each week for 6weeks. Each phone call is expected to last around 1 hour with flexibility to be shorter or longer. The calls will be unstructured and designed simply to engage in conversation with the participant. The length of the phone calls, days and times will be recorded by the volunteer along with a short journal entry describing the conversation topics and any information that stood out to the volunteer. If the stroke survivor and student volunteer wish to speak more than the designated one call a week, that will be allowed if both parties agree. The same student volunteer will conduct all six sessions

SUMMARY:
The purpose of this study is to see the impact of social visits, through weekly phone calls, on quality of life and health outcomes of depression, anxiety, loneliness, and self-rated health for adults who have experienced an ischemic or hemorrhagic stroke and to determine the benefit of these conversations on the student volunteer's perspective of adults who have survived a stroke

ELIGIBILITY:
Inclusion Criteria:

* have a UCLA short form score of 4 or higher
* can read, write, and speak English
* have had an ischemic or hemorrhagic stroke is the past year
* have a telephone and are available for weekly phone calls
* provide informed consent agreeing to be contacted by the volunteers

Exclusion Criteria:

* reside outside of the home
* have Electronic Health Record documentation of Aphasia
* Montreal Cognitive Assessment score of <9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of participants who enrolled in the study | post intervention (6 weeks from start of intervention)
Feasibility as assessed by the number of participants who completed all 6 phone calls | post intervention (6 weeks from start of intervention)
Feasibility as assessed by the number of participants who completed all the assessments | post intervention (6 weeks from start of intervention)

SECONDARY OUTCOMES:
Change in loneliness as assessed by the University of California, Los Angeles (UCLA) Loneliness Scale | Baseline, post intervention (6 weeks from start of intervention)
  This is a 20 item questionnaire, each one is scored form 1(never) to 4(always). Scores for questions 1,5,6,9,10,15,16,19 and 20 are reversed(i.e. 1=4,2=3,3=2,4=1)and the scores for each item is then summed together, higher number indicating more loneliness
Change in depression as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, post intervention (6 weeks from start of intervention)
  This is a 20 item questionnaire, each item is scored from 0(rarely or none of the time)-3 (most or all of the time) with a possible range of scores from 0-60 a higher score indicating more depression
Change in anxiety as assessed by the Generalized Anxiety Disorder 7 Scale (GAD 7) | Baseline, post intervention (6 weeks from start of intervention)
  This is a 7 item questionnaire, each is scored from 0(not at all) to 3(nearly every day) a higher number indicating more anxiety
Change in social support as assessed by the Duke Social Support Index (DSSI) Scale | Baseline, post intervention (6 weeks from start of intervention)
  This is a 10 item questionnaire and each is scored from 1-3,with a maximum score of 30 and higher score indicating higher levels of support
Change in resilience as assessed by the brief resilience scale | Baseline, post intervention (6 weeks from start of intervention)
  This is a 6 item questionnaire and each is measured from 1(strongly disagree)-5(strongly agree) for maximum score of 30 a higher score indicating greater resilience to stressful events
Change in pain as assessed by the Brief Pain Inventory Short Form | Baseline, post intervention (6 weeks from start of intervention)
  This questionnaire has 2 subscales :
  The first subscale is the pain severity subscale which consists of 4 questions and each are scored from 0(no pain)-10(severe pain), a higher number indicating more pain
  The second subscale is the pain interference score and it contains 7 items and each is scored from 0(does not interfere)-10(completely interferes) a higher number indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Beauchamp, PhD, RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No